CLINICAL TRIAL: NCT03181555
Title: Pilot Study: Identification of a Multi-omic Predictive Signature for Preterm Birth in Obese African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Principal Investigator, Mary Ann Faucher, Associate Professor, Baylor University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 916539
Record Dates: First submitted 2016-12-09; First posted 2017-06-09 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: PREG1; Obesity
Keywords: Pregnant; Obese; Omic
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Masking Description: No masking. A convenience sample of pregnant AA women will be recruited based on race/ethnicity and body mass index.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnant Obese African American Women (Other): Exploratory
  Interventions: Other: Exploratory

INTERVENTIONS:
Other: Exploratory

SUMMARY:
1. Determine if the stool or vaginal microbiome and urinary metabolite profiles in a pregnant obese population of African American women differ from their pregnant non-obese counterparts
2. Determine if the stool or vaginal microbiome and urinary metabolite profiles vary by class of obesity and magnitude of excess weight gain in this population of pregnant African-American women.
3. Assess the ability of the stool, vaginal microbiome, or metabolites, or the combination of all biomarkers as predictors of preterm birth (PTB) and onset of labor.
4. Determine if any dietary or clinical variables are correlated with changes in the microbiome or urinary metabolites or modify their association with PTB

DETAILED DESCRIPTION:
This is an exploratory pilot study to determine the omic footprint in pregnant AA women and then compare difference between obese and non-obese pregnant AA women and comparisons by class of obesity. Variations in the omic findings (vaginal and gut microbiome and urinary metabolites) will be assessed by dietary findings and by variations in gestational weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 or older English Speaking Access to internet- The dietary assessment for this study is The Automated Self-Administered 24-hour Recall (ASA24-2014), a web-based instrument developed by researchers at the National Cancer Institute (NCI).

Exclusion Criteria:

- 1. History of preterm birth and taking progesterone. Progesterone may influence the microbiota and metabolites so therefore these women will not be eligible for the study. However, if the women fit other inclusion criteria and have a history of preterm birth but are not on progesterone they will be eligible for enrollment 2. History of antibiotic use in the last month (includes pre-biotics and probiotics). These medications will change the baseline microbiota.

3. History of chronic disease on medications

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
1. Differences in vaginal and gut microbiome and urinary metabolites profile between obese and nonobese pregnant AA women | 27-28 weeks to 39 weeks of pregnancy
  The vaginal and gut microbiome and urine metabolites in obese women AA women will be compared with non-obese pregnant AA women. This comparison will be investigated by diet and gestational weight gain

SECONDARY OUTCOMES:
Differences in vaginal and gut microbiome and urinary metabolites profile between by class of obesity in pregnant AA women | 27-28 weeks to 39 weeks of pregnancy
  The vaginal and gut microbiome and urine metabolites in obese women AA women will be compared by class of obesity. This comparison will be investigated by diet and gestational weight gain

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Faucher, PhD, Principal Investigator — Baylor University
Locations (1):
- MacArthur OB/GYN, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No